CLINICAL TRIAL: NCT03607591
Title: Efficacy of High Frequency (15Hz) Repetitive Transcranial Magnetic Stimulation of Left Dorsolateral Prefrontal Cortex in Decreasing Intake in Patients With Cocaine Use Disorder: Study Protocol for a Randomized Placebo Controlled Trial
Brief Title: Efficacy of Repetitive Transcranial Magnetic Stimulation in Reducing Cocaine Intake in Addicted Patients
Acronym: MagneTox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Antonello Grippo, Medical Doctor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEAVC SPE 16.309
Record Dates: First submitted 2018-04-13; First posted 2018-07-31 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Cocaine Use Disorder
Keywords: rTMS; Craving; Mood and cognitive behavior; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS group (Active Comparator): One daily session: active 15Hz frequency, pulse intensity 100% of the rTMS, 60 pulses per train, inter-train pause of 15 sec, 40 stimulation trains for a total of 2400 pulses in 13 min of stimulation). 15 sessions (3 weeks of 5 consecutive daily sessions and 2 days of rest)
  Interventions: Other: rTMS
- Placebo rTMS group (Placebo Comparator): One daily session: inactive 15Hz frequency, pulse intensity 100% of the rTMS, 60 pulses per train, inter-train pause of 15 sec, 40 stimulation trains for a total of 2400 pulses in 13 min of stimulation). 15 sessions (3 weeks of 5 consecutive daily sessions and 2 days of rest)
  Interventions: Other: rTMS

INTERVENTIONS:
Other: rTMS — rTMS is a non-invasive and safe brain stimulation technique, that uses a magnetic pulse, administrated through a coil, set on the DLPFC

SUMMARY:
The study evaluates the efficacy of 3 weeks of repetitive transcranial magnetic stimulation (rTMS), 5 sessions/weekly, in reducing cocaine consumption immediately after and within the 8 weeks following the treatment in addicted patients with cocaine use disorders (CUD) versus placebo.

DETAILED DESCRIPTION:
40 patients are expected and randomized in two groups: 20 patients with active rTMS and 20 with placebo rTMS.

Visit 1: 15 days (3 weeks of 5 consecutive daily sessions and 2 days of rest) 15Hz rTMS is performed during the following days in addition to a biweekly urine drug test and VAS evaluation.

Visit 2: Changes from baseline to week 8 in cocaine intake. Evaluation of craving and of other assessments like mood and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between 18 and 65 years of age
* patients who meet the criteria for CUD reported in the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V)
* positivity to cocaine use, determined via an urine drug test
* patients who are able to provide a written informed consent, after being notified about the treatment and the study protocol

Exclusion Criteria:

* major depression disorder, schizophrenia, bipolar disorder or other psychosis that meet the diagnostic criteria of the DSM-V
* illiteracy or cognitive impairment disorders
* women who are pregnant or lactating
* other medical diseases that contraindicate rTMS treatment such as epilepsy
* presence of devices, i.e. pace-makers or cochlear prosthesis
* previous rTMS treatments in order to avoid confounding factors
* patients who can not provide the written informed consent
* DSM-V substance use disorders other than CUD. Only tobacco smoke is allowed to be recruited in the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Cocaine intake | 8 weeks following the treatment
  Baseline was defined as cocaine consumption before randomization (visit 0). Baseline will be determined using an urine drug test.Changes from baseline to week 8 in cocaine intake

SECONDARY OUTCOMES:
Craving first measure | 8 weeks following the treatment
  Baseline will be determined using the Visual Analogic Scale (VAS) that is a ordinal scale ranging from 0 to 10. being 0 no craving and 10 maximum craving. Changes from baseline to 8 week
Craving second measure | 8 weeks following the treatment
  Baseline will be assessed using Cocaine Craving Questionnaire (CCQ), that is a ordinal scale ranging from 0 and 45, being 0 no craving and 45 maximum craving.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lolli F, Salimova M, Scarpino M, Lanzo G, Cossu C, Bastianelli M, Occupati B, Gori F, Del Vecchio A, Ercolini A, Pascolo S, Cimino V, Meneghin N, Fierini F, D'Anna G, Innocenti M, Ballerini A, Pallanti S, Grippo A, Mannaioni G. A randomised, double-blind, sham-controlled study of left prefrontal cortex 15 Hz repetitive transcranial magnetic stimulation in cocaine consumption and craving. PLoS One. 2021 Nov 16;16(11):e0259860. doi: 10.1371/journal.pone.0259860. eCollection 2021. PMID 34784373